CLINICAL TRIAL: NCT04122495
Title: Treatment of Upper and Lower Respiratory Tract Infections in Young Children Using Probiotic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Beijing Scitop Bio-Tech Shareholding Co.Ltd. (Unknown)
Responsible Party: Principal Investigator, Min-Tze LIONG, Prof. (Clinical Professor), Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USM/JEPEM/19030177
Record Dates: First submitted 2019-09-30; First posted 2019-10-10 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Infection (for Example, Pneumonia, Bronchitis)
Keywords: probiotic; respiratory tract infections; Bifidobacterium; children
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia; Bronchitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Bifidobacterium lactis M8 at 10 log CFU/day for 4 weeks
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Intervention consists of daily administration of 1g of maltodextrin, administered daily for 4-weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Oral administration of B. lactis M8 at 10 log CFU/day for 4-weeks
  Other Names: Bifidobacterium lactis M8
  Arms: Probiotic
Dietary Supplement: Placebo — Oral administration of maltodextrin daily for 4-weeks
  Arms: Placebo

SUMMARY:
This project aims to study the benefits of probiotics namely Bifidobacterium lactis M8 in treatment of upper and lower respiratory tract infections in young children, which are found common among children in Malaysia aged from 0-24 months.

DETAILED DESCRIPTION:
Respiratory illnesses are the most common acute diseases in children where no virtually effective treatments or prophylaxes are available for these infections. Probiotics on the other hand have gained increasing evidences as an effective therapy in preventing respiratory tract infections. While the precise mechanisms of using probiotics in management of respiratory infections are largely unknown, speculations include: probiotics compete against pathogens; increase the barrier function in respiratory epithelium; immunostimulatory effects by enhancing cellular immunity with increased activity of natural killer cells and macrophages in airways. Hence, probiotics may offer safe means of reducing the risk of early respiratory related illnesses, common cold and antibiotic use, and the risk of recurrent respiratory infections, thereby represent a simple, safe, effective, available and affordable method for preventing respiratory infections in children.

Among the various types of probiotics, Bifidobacterium is one of the best-known probiotic genus in the world, and it is widely applied in the dairy industry as a probiotic. Evidences from more than 100 scientific publications based on in vitro, in vivo, and clinical studies and long consumption history support the safety and health benefits of Bifidobacterium strains. The ingestion of yogurt fortified with B. longum reduced harmful bacteria such as Enterobacteriaceae, Streptococcus and C. perfringens, while at the same time alter the microbiota gut profile of volunteers with a significant increase of beneficial microbes Bifidobacterium and Lactobacillus species. Additionally, putrefactive substances in the intestinal environment were also reduced in the presence of the probiotic supplement. Such findings suggest that Bifidobacterium strains are safe and could be used further to evaluate its effect in preventing diarrhea and/or respiratory-related illness prevalence in young children.

Bifidobacterium lactis M8 was isolated from breast milk samples collected from healthy woman in China. M8 was selected as it was the best among 857 other strains with excellent tolerance to gastric acid, intestinal fluid and bile salt of the digestive system. M8 is manufactured under a ISO9001 and ISO22000 certified manufacturing plant (JinHua YinHe Biological Technology Co. Ltd., China). M8 does not contain any porcine or bovine ingredients and has obtained the HALAL certification from ARA HALAL Development Services Center Inc. (ARA), which is recognized by JAKIM, Malaysia.

M8 is incorporated and sold in the market of China, Taiwan and Singapore in a variety of products, ranging from dairy (yoghurt and fermented milk). The product M8 contains good bacteria Bifidobacterium lactis M8 and primarily maltodextrin as carrier while placebo contains primarily maltodextrin. Sachets of products containing probiotic M8 and placebo appear as light yellow powder. Both M8 and placebo products are kept at storage temperature range below 30oC according to the condition recommended by the manufacturer.

A total number of 120 respiratory-related hospitalized children from age 0-24 months old will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* young children aged 1-24 month, admitted to hospital for having respiratory diseases.
* Willing to commit throughout the experiment

Exclusion Criteria:

* Long term medication due to certain severe illness
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization in young children with respiratory tract infections upon administration of B. lactis M8 | 4-weeks
  Differences in duration of hospitalization in young children with respiratory tract infections upon administration of B. lactis M8 at 10 log CFU/day compared to placebo

SECONDARY OUTCOMES:
Clinical symptoms in young children with respiratory tract infections upon administration of B. lactis M8 as assessed using the Monthly Health Questionnaire (as used in ClinicalTrials.gov (identifier number NCT02434042). | 4-weeks
  Differences in number of days and duration of symptoms of young children with respiratory tract infections upon administration of B. lactis M8 at 10 log CFU/day compared to placebo
Clinical symptoms in young children with respiratory tract infections upon administration of B. lactis M8 as assessed using the Monthly Gastrointestinal Questionnaire as used in ClinicalTrials.gov (identifier number NCT02434042). | 4-weeks
  Differences in number of days and duration of symptoms of young children with gastrointestinal infections upon administration of B. lactis M8 at 10 log CFU/day compared to placebo
Microbiota profiles of saliva and fecal samples in young children with respiratory tract infections upon administration of B. lactis M8 as assessed via pyrosequencing | 4-weeks
  Differences in microbiota abundance of saliva and fecal sample in young children with respiratory tract infections upon administration of B. lactis M8 at 10 log CFU/day compared to placebo
Concentrations of proteins in saliva and fecal samples in young children with respiratory tract infections upon administration of B. lactis M8 as assessed via biochemical tests | 4-weeks
  Differences in concentrations of protein such as interleukins (IL-10, IL-4, IL-6, TNF-alpha, IFN-gamma) in saliva (ug/mL) and fecal (ug/mg) sample in young children with with respiratory tract infections upon administration of B. lactis M8 at 10 log CFU/day compared to placebo
Gene expressions for inflammation and immunity from saliva and fecal samples in young children with respiratory tract infections upon administration of B. lactis M8 as assessed via real time PCR | 4-weeks
  Differences in gene expressions for inflammation (IL-10, IL-4, IL-6, TNF-alpha, IFN-gamma), immunity (T-cell and B-cell) in unit of fold change or delta-delta CT values, of saliva and fecal sample in young children with respiratory tract infections upon administration of B. lactis M8 at 10 log CFU/day compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Min Tze Liong, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital USM, Kubang Kerian, Kelantan, Malaysia

REFERENCES:
- [Derived] Mageswary MU, Ang XY, Lee BK, Chung YF, Azhar SNA, Hamid IJA, Bakar HA, Roslan NS, Liu X, Kang X, Dai L, Sreenivasan S, Taib F, Zhang H, Liong MT. Probiotic Bifidobacterium lactis Probio-M8 treated and prevented acute RTI, reduced antibiotic use and hospital stay in hospitalized young children: a randomized, double-blind, placebo-controlled study. Eur J Nutr. 2022 Apr;61(3):1679-1691. doi: 10.1007/s00394-021-02689-8. Epub 2021 Nov 26. PMID 34825264